CLINICAL TRIAL: NCT05526469
Title: Ultrasound-Guided Single Shoot Serratus Anterior Plane Block Versus Erector Spinae Plane Block as Novel Techniques for Post-Thoracotomy Pain Control in Pediatric Cardiac Surgery and Its Effect in Ultra-Fast Track Recovery: A Prospective Randomized Trial
Brief Title: Ultrasound-Guided Serratus Anterior Plane Block Versus Erector Spinae Plane Block in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Akram Mohamed Mohamed Amer, MD, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 110/ 2022
Record Dates: First submitted 2022-08-01; First posted 2022-09-02 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease
Keywords: Pediatric; Cardiac surgery; Ultrasound; Serratus anterior plane block; Erector spinae plan block
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group serratus anterior plane (SAP) (Active Comparator): patients will receive ultrasound guided single shot serratus anterior plane block with 0.5 ml/kg bupivacaine 0.25%
  Interventions: Procedure: Serratus anterior plane block; Drug: Bupivacaine 0.25% Injectable Solution
- Group erector spinae plane (ESP) (Active Comparator): patients will receive ultrasound guided single shot erector spinae plane block with 0.5 ml/kg bupivacaine 0.25%
  Interventions: Procedure: erector spinae plane blocks; Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Procedure: Serratus anterior plane block — patients in this group will receive ultrasound guided single shot serratus anterior plane block for pain control intra and postoperative
  Arms: Group serratus anterior plane (SAP)
Procedure: erector spinae plane blocks — patients in this group will receive ultrasound guided single shot erector spinae plane block for pain control intra and postoperative
  Arms: Group erector spinae plane (ESP)
Drug: Bupivacaine 0.25% Injectable Solution — Patients in both group will receive 0.5 ml/kg bupivacaine 0.25% injected locally in the muscle plane

SUMMARY:
Background and Objectives: Opioid based analgesia is the main used technique in pediatric cardiac surgery which preclude fast-track recovery. Ultrasound guided regional fascial plane blocks are used recently in many pediatric surgical procedure with excellent outcomes and very low rate of complication. The investigators will compare ultrasound guided serratus anterior plane block and erector spinae plane block in pediatric cardiac surgical procedure through thoracotomy approach regarding effectiveness of postoperative analgesia, incidence of complications and effect in ultrafast track recovery.

Methods: The investigators will enroll 64 pediatric patients aged from 6 months to 10 years undergoing cardiac surgical procedure through thoracotomy approach either with or without cardiopulmonary bypass in this prospective randomized study. After induction of general anesthesia, the patients will be randomly assigned into 2 groups based regional fascial plane block given (SAP group will receive ultrasound guided single shot serratus anterior plane block and ESP group will receive ultrasound guided single shot erector spinae plane block). The effectiveness of postoperative analgesia using FLACC pain score will be recorded as the primary outcome while total consumption of analgesics, the time for rescue analgesia, incidence of complications, and incidence of need for re-intubation will be recorded as the secondary outcomes.

DETAILED DESCRIPTION:
INTRODUCTION:

Pain control in pediatric cardiac surgery is an area of great interest with opioid based analgesia is the mainstay used technique. Use of high doses of opioid usually preclude early/ultrafast track recovery and extubation in operating room (OR). The benefits of ultrafast track recovery include shorter intensive care unit (ICU) and hospital stay, lower incidence of postoperative complications, reduce occurrence of ventilator induced complications and infection, with better hemodynamics.

With the era of regional anesthetic techniques, there is an increasing need to use a novel techniques of fascial plane block in pain control post cardiac surgery especially the use of neuraxial blocks carry a great risk of spinal hematoma with use of high doses of heparin.

Ultrasound (U/S) guided serratus anterior plane block (SAPB) and erector spinae plane block (ESPB) are used recently in many thoracic, breast and chest wall surgeries with high success rate, low incidence of complications, and solid pain control with many studies demonstrated superior efficacy in comparison to classic analgesic techniques. The use of SAPB and ESPB in cardiac surgery in general and pediatric cardiac surgery are very limited. Both techniques have been used in pediatric cardiac surgical procedures and provided a promising effect as a simple, safe, and effective postoperative analgesic techniques.

The current study will compare the 2 novel fascial plane blocks -SAPB and ESPB- in pain control and effectiveness for ultrafast track recovery in pediatric cardiac patients undergoing cardiac surgical procedure through thoracotomy approach with or without cardiopulmonary bypass (CBP). The primary outcome will be the effectiveness of postoperative analgesia using FLACC (Face, Leg, Activity, Cry and Consolability) pain score and the secondary outcome will be the total consumption of postoperative analgesics, the time for first rescue analgesia, incidence of complications up to 24 hours, and incidence of need for re-intubation in the first 6 hours.

AIM/ OBJECTIVES:

1. To compare the effectiveness of postoperative analgesia using FLACC pain score in patients receiving SAP block versus ESP block in pediatric cardiac patients undergoing cardiac surgical procedure through thoracotomy approach (primary outcome).
2. To determine the effect of SAP block on total consumption of postoperative analgesics, the time for first rescue analgesia, incidence of complications up to 24 hours, and incidence of need for re-intubation in the first 6 hours as compared to ESP block (secondary outcome).

METHODOLOGY:

The study will be conducted at Ain Shams University Hospitals after ethical committee approval and obtaining an informed written consent from patients' guardian.

* Type of Study; Randomized single blinded clinical trial.
* Study Setting; Pediatric cardiac surgery operating theatre in Ain shams university hospital, Cairo, Egypt.
* Study Period; The study will be started immediately after ethical committee approval starting August 2022 aiming to be completed within 6 months.
* Study Population

  * Inclusion Criteria: The patients will be of ASA (American Society of Anesthesiology) physical status II-III, aged between 6 months and 10 years old, of both sexes, and undergoing cardiac surgical procedure through thoracotomy approach either with or without cardiopulmonary bypass e.g. atrial septal defect (ASD) closure, patent ductus arteriosus (PDA) ligation, and aortic coarctation repair.
  * Exclusion Criteria: included patients weight less than 5 kg, coagulopathy, previous cardiac surgery, emergency procedure, previous thoracotomy or sternotomy, surgery through sternotomy incision, patients with complex surgical repair, and patients need postoperative mechanical ventilation. Other exclusion criteria included hypersensitivity to local anesthetics, infection at site of block injection, and parent or guardian refusal.
* Sampling Method; Based on the block will be performed, patients will be randomly and evenly assigned to one of two groups (32 patients each) using a computer-generated list: Group SAP (serratus anterior plane) and group ESP (erector spinae plane).

Group SAP: patients will receive ultrasound guided single shot serratus anterior plane block with 0.5 ml/kg bupivacaine 0.25%.

Group ESP: patients will receive ultrasound guided single shot erector spinae plane block with 0.5 ml/kg bupivacaine 0.25%.

* Sample Size; This is a pilot clinical trial with no similar previous studies. The primary outcome is to compare the mean score of the Pain scale between ESP and SAP at different periods after extubation. Assuming large effect size of 0.8, A sample size of at least 32 cases per group - totaling 64 cases in two groups - achieves a power of 80% to detect a large effect size of 0.8 comparing the mean pain scores of the two groups using two independent samples t-test with level of confidence of 0.05. Sample size is inflated by 20% to compensate for dropouts.
* Ethical Considerations; After acquiring local medical ethics committee approval and informed written consent from the parent or guardian, we will enroll 64 patients in this study.
* Study Tools AND/ OR Study Procedures AND/OR Study Interventions; All patients will be assessed and prepared preoperatively according to local hospital protocol. All patients will be premedicated with IV Midazolam 0.1mg/kg 5 minutes before surgery (maximum of 2.5 mg). Routine monitoring with 5-lead ECG, non-invasive blood pressure and pulse oximetry will be instituted, then anesthesia will be induced with IV propofol 2-3mg/kg, fentanyl 2mcg/kg, and cisatracurium 0.2 mg/kg, to facilitate endotracheal intubation. Sevoflurane (1%-2%) in 30-50% oxygen in air mixture will be used for maintenance of anesthesia. Cisatracurium infusion 2mcg/kg/min will be started after insertion of CVP line and will be discontinued 30 min before skin closure. After intubation, all children will be mechanically ventilated with volume control ventilation using 7-10 mL/kg tidal volume, maintaining end-tidal carbon dioxide tension around 30-35 mmHg. Arterial line and central venous catheter will be inserted to all patients. One of the 2 regional nerve blocks (SAP, or ESP) will be performed with ultrasound guidance per group allocation. The blocks will be performed with aseptic precautions using an 8 to13 megahertz (MHz) linear probe (Philips®) in a sterile cover with sterile jelly and a 22-gauge 50 mm echogenic block needle (SonoPlex® PAJUNK® , Germany).

Technique of SAP block; while the patient in the lateral position with the surgical/block side upward, the ultrasound transducers will be placed in a sagittal plane over the midclavicular area of the thoracic wall then the ribs will be counted till the 5th rib will be identified in the midaxillary line. The following muscular layers will be recognized from superficial to deep layers; latissimus dorsi then serratus anterior muscles. The needle will be introduced from caudal to cranial direction with in-plane technique as related to the ultrasound probe targeting the plane between the two muscles. Under real lime U/S guidance, the local anesthetic solution will be injected after negative aspiration to blood or air with making sure to visualize the plane of separation between the two muscles.

Technique of ESP block; while the patient in the lateral position with the surgical/block side upward, the ultrasound transducers will be placed in a parasagittal plane 2-3 cm away from the dorsal midline at the level of 5th thoracic vertebrae. Sliding the transducer medially till identifying the transverse process which appear as flat acoustic shadow (the ribs appears as rounded acoustic shadows more laterally) with an interceding hyperechoic pleural line. The following muscular layers will be recognized from superficial to deep layers; trapezius, rhomboid, then erector spinae muscles. The needle will be introduced either cranio-caudal or caudo-cranial direction with in-plane technique as related to the ultrasound probe targeting the plane between the erector spinae muscle and transverse process of T5. Under real lime U/S guidance, the local anesthetic solution will be injected after negative aspiration to blood or air with making sure to visualize the plane of separation under the erector spinae muscle.

Any complications related to the block given will be recorded including hematoma, intravascular injection, and allergic reactions. The duration of performing the block will be also recorded. Intraoperative hemodynamic parameters will be recorded including heart rate (HR), systolic blood pressure (SBP), mean arterial pressure (MAP), respiratory rate (RR), and peripheral oxygen saturation (SPO2) at the following intervals; baseline before induction of anesthesia, just before skin incision, after skin incision, 15 min after skin incision, at the end of surgery, and after extubation. Total doses of intraoperative opioids including fentanyl and or morphine will be calculated and recorded.

After skin closure inhalational anesthesia will be discontinued and reversal of muscle relaxant after returning of spontaneous breathing will be acquired. Tracheal extubation will be performed after ensuring adequate tidal volume, respiratory rate along with hemodynamic stability, normothermia, normal blood gases parameters, and the patient is fully conscious. After extubation and ensuring hemodynamic stability, the patient will be transferred to ICU fully monitored and connected to oxygen simple face mask 6 L/min.

Pain assessment will be done using the FLACC pain scale score at the following intervals; immediate post-extubation, every 1 hour for the 1st 6 hours postoperatively then every 2 hours for the next 6 hours then every 4 hours till 24 hours postoperatively. Rescue analgesic will be used if FLACC pain scale score is 4 or more according to hospital protocol. Time of the 1st postoperative rescue analgesia will be recorded, also total doses of analgesic given will be recorded.

Postoperative hemodynamic parameters will be recorded including HR, SBP, MAP, RR, and SPO2 at the following intervals; hourly for the 1st 6 hours postoperatively then every 2 hours for the next 6 hours.

Need for tracheal re-intubation within 6 hours from recovery will be considered as failed ultrafast trach recovery and will be recorded. Length of stay in ICU will be recorded.

The data during surgery and after surgery will be collected by the resident anesthetist not involved in the study.

* Statistical Analysis; Numerical data are presented as the mean (standard deviation) or median (range) while categorical data are presented as the number of cases (percentage). Between-group comparisons of numerical variables will be performed by the independent sample T-test, or Mann-Whitney test as appropriate, while those of categorical variables will be performed by the Chi-square test. For all tests, a P (probability) value < 0.05 will be considered statistically significant.
* Statistical Package; The data collected will be analyzed with statistical program SPSS (version 22.0 Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II-III.
* Age between 6 months and 10 years old,
* of both sexes,
* undergoing cardiac surgical procedure through thoracotomy approach either with or without cardiopulmonary bypass e.g. ASD closure, PDA ligation, and aortic coarctation repair.

Exclusion Criteria:

* Patients weight less than 5 kg,
* Patients with coagulopathy,
* previous cardiac surgery,
* emergency procedure,
* previous thoracotomy or sternotomy,
* surgery through sternotomy incision,
* patients with complex surgical repair,
* patients need postoperative mechanical ventilation.
* hypersensitivity to local anesthetics,
* infection at site of block injection,
* parent or guardian refusal.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of postoperative analgesia | 6 months
  We will test the effect of serratus anterior plane block in adequacy of postoperative analgesia (using FLACC pain scale "from 0 to 10") compared to erector spinae plane block

SECONDARY OUTCOMES:
Incidence of complications | 6 months
  We will test the effect of serratus anterior plane block in incidence of complications (including hematoma, intravascular injection, and allergic reactions "measured as a percentage") compared to erector spinae plane block
Tracheal re-intubation | 6 months
  We will test the effect of serratus anterior plane block in incidence of tracheal re-intubation within 6 hours postoperative (measured as a percentage) compared to erector spinae plane block
Length of ICU stay | 6 months
  We will test the effect of serratus anterior plane block in length of ICU stay (measured in hours) compared to erector spinae plane block

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university- faculty of medicine- department of anesthesia, intensive care and pain management, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through the study may be provided to qualified researchers with academic interest in pediatric cardiac anesthesia. Data shared will be coded, with no patient health information included.
Supporting Information: Study Protocol, CSR
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. For more information or to submit a request, please contact akram.amer@med.asu.edu.eg